CLINICAL TRIAL: NCT01366365
Title: A Phase 1 Randomized, Double-Blind, Placebo Controlled Parallel Group Study of the Pharmacokinetics, Safety and Tolerability of Methylnaltrexone Bromide Administered as Single and Multiple Intravenous Doses to Healthy Adults and Elderly Male and Female Subjects
Brief Title: Study of Pharmacokinetics, Safety and Tolerability of Intravenous Methylnaltrexone Bromide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Tage Ramakrishna, MD, Progenics Pharmaceuticals, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MNTX 1303
Record Dates: First submitted 2011-05-27; First posted 2011-06-06 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Healthy Adults
MeSH Terms: interventions — methylnaltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): IV methylnaltrexone (MNTX)
  Interventions: Drug: methylnaltrexone
- Arm 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: methylnaltrexone
  Arms: Arm 1
Drug: placebo
  Arms: Arm 2

SUMMARY:
This double-blind, randomized, two-cohort, placebo-controlled, parallel group study characterized the pharmacokinetics, safety, and tolerability of MNTX following single doses and at steady-state during multiple dosing and assessed the effects of aging on the pharmacokinetics, safety and tolerability of MNTX.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Males and females who were between the ages of 18 and 45 years and healthy males and females who were 65 years of age and older.
2. Subjects who were non-smokers
3. Subjects with body weights within range of 70-100 kg (154-220 lbs).

Exclusion Criteria:

1. Subjects who had previously been exposed to MNTX
2. Subjects with a history of vasovagal episodes or fainting within the past five years
3. Subjects with a history of psychiatric or neurologic disorder
4. Subjects with a history of narrow-angle glaucoma or intraocular hypertension
5. Subjects who had tested positive for hepatitis B surface antigen, IgM hepatitis B core antibody, hepatitis C antibody, or HIV
6. Subjects who have had a diagnosis of alcohol or substance dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-10; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Clearance of MNTX | 7 days
  Evaluate the PK of MNTX in healthy adult and healthy elderly male and female human subjects following MNTX administration as a single IV dose, and at steady state during multiple IV doses

SECONDARY OUTCOMES:
Half-life of MNTX | 7 days
  Evaluate the PK of MNTX in healthy adult and healthy elderly male and female human subjects following MNTX administration as a single IV dose, and at steady state during multiple IV doses
Volume of distribution of MNTX | 7 days
  Evaluate the PK of MNTX in healthy adult and healthy elderly male and female human subjects following MNTX administration as a single IV dose, and at steady state during multiple IV doses
Area under the plasma concentration (AUC) of MNTX | 7 days
  Evaluate the PK of MNTX in healthy adult and healthy elderly male and female human subjects following MNTX administration as a single IV dose, and at steady state during multiple IV doses
Number of Subjects with Adverse Events | 7 days
  Safety and tolerability of MNTX in healthy adult and healthy elderly male and female human subjects following MNTX administration as a single IV dose, and at steady state during multiple IV doses

CONTACTS AND LOCATIONS:
Overall Officials: Tage Ramakrishna, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States